CLINICAL TRIAL: NCT05847036
Title: Profiles of Urinary Tract Infections in General Practice : a Prospective Multicentre Cohort Study
Brief Title: Profiles of Urinary Tract Infections in General Practice
Acronym: PODIUM
Status: Recruiting | Type: Observational
Sponsor: CNGE Conseil (Other)
Responsible Party: Sponsor
Other Study IDs: CNGE-2021-05
Record Dates: First submitted 2023-04-07; First posted 2023-05-06 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urinary tract infections (UTIs) are one of the most common bacterial infections managed in general practice: they are the 2nd site of community-acquired bacterial infection after respiratory infections (4-6 million consultations per year in France).

UTIs represent 15% of total antibiotic prescriptions in France. Antibiotics recommended for UTIs, except for cystitis, are considered as "critical" (highly generating bacterial resistances). UTIs are a potential source of antibiotic resistance: often inappropriate antibiotic prescriptions, evolution of the resistance profiles of the bacteria involved, emergence of multi-resistant strains.

The first hypothesis is that there are other profiles of clinical UTI situations in general practice than typical cystitis or pyelonephritis, including intermediate forms.

The second hypothesis is that these intermediate forms of UTI are subject to longer durations of antibiotherapy, and that probable explanatory factors need to be identified.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are one of the most common bacterial infections managed in general practice: they are the 2nd site of community-acquired bacterial infection after respiratory infections (4-6 million consultations per year in France).

UTIs represent 15% of total antibiotic prescriptions in France. Antibiotics recommended for UTIs, except for cystitis, are considered as "critical" (highly generating bacterial resistances). UTIs are a potential source of antibiotic resistance: often inappropriate antibiotic prescriptions, evolution of the resistance profiles of the bacteria involved, emergence of multi-resistant strains.

Current guidelines classify UTIs as "uncomplicated UTI" (cystitis and pyelonephritis) and "UTI at risk of complication" (cystitis, pyelonephritis and male UTI) [1-2]. However, in primary care, pathologies are diagnosed at an early stage: the clinical signs usually described by scientific societies are not always all found, and the descriptions are not always adapted to the realities encountered in general practice [3-6]. Some clinical situations do not fit into the systematic categories of the guidelines, with "intermediate" forms (such as pain in the lumbar fossae without fever "cysphritis" or other atypical presentations) [3]. The current literature in general practice highlights these issues: the need for prospective cohorts in real-life practice to identify these profiles and develop more appropriate guidelines [3-6]. Treatment for these intermediate forms is not obvious and is often empirical: potentially longer antibiotherapies, with possible worsening of antibiotic resistance [7].

The first hypothesis is that there are other profiles of clinical UTI situations in general practice than typical cystitis or pyelonephritis, including intermediate forms.

The second hypothesis is that these intermediate forms of UTI are subject to longer durations of antibiotherapy, and that probable explanatory factors need to be identified.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years old
* Patient presenting one or more of the following clinical signs suggestive of urinary tract infection in general practice consultation:

  * fever (temperature > 38°C)
  * chills, sweats
  * burning urination
  * urinary urgency
  * pollakiuria
  * dysuria
  * lumbar and/or pelvic pain
  * abnormal urine appearance: cloudy, malodorous, macroscopic haematuria
  * absence of leucorrhoea
  * specifically in people > 70 years old:

    * recent onset urinary incontinence
    * sudden confusion
    * bladder globe
* Positive urine dipstick and/or positive Cytobacteriological Examination of Urine (CBEU)
* Patient affiliated with the French National Health Insurance or beneficiary of such a scheme.
* Patient's oral non-opposition of participation in the study after receiving complete information about the protocol

Non-inclusion Criteria:

* Patient < 18 years old
* Declared pregnancy
* Patient with indwelling urinary catheter
* Patient with functional or organic abnormality of the urinary tract
* Patient with known severe immunodeficiency (HIV+ with CD4 count < 200/mm3, organ transplant, bone marrow transplant, patient on immunosuppressants, cirrhosis)
* Patient with known severe chronic renal failure (clearance < 30 mL/min)
* Patient previously treated with an antibiotic (for an other reason than a urinary tract infection and/or treatment failure of the urinary tract infection) in the past month before the inclusion consultation
* Patient speaking little or no French
* Patient with severe cognitive impairment
* Patient with life expectancy < 3 months
* Patient under legal protection, inability to give an oral non-opposition
* Patient with severity criteria justifying hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients consulting in general practice for suspected urinary tract infection
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the number of homogeneous profiles of patients with UTI in general practice and their characteristics using clinico-bacteriological indicators. | At Day 14 after the end of the Antiobiotic treatment
  The primary outcome will be the rate and the clinical-bacteriological characteristics of the identified profiles of patients with UTI in general practice

SECONDARY OUTCOMES:
For general practioners' practices: | At Day 0, at Day 14 after the end of the treatment and between Day 0 and Day14 after the end of the treatment
  Percentage of cytobacteriological examination of urine (CBEUs) prescribed
  * Number and type of additional examinations prescribed
  * Percentage of antibiotics prescribed, therapeutic class chosen, duration (in ordinal categories), posology
For short-term evolutionary trajectories: | At Day 0, at Day 14 after the end of the treatment and between Day 0 and Day 14 after the end of the treatment
  Number of consultations (in general practice or other specialty) and reasons
  * Number of emergency department visits
  * Number of unscheduled hospitalizations related to UTI
For short-term evolutionary trajectories: | At Day 14 after the end of the treatment
  Percentage of patients with worsening, stability or recovery of their symptoms as final condition (based on clinical assessment by GPs during a consultation at day 14)
For the factors associated with the prescription of antibiotics: | At Day 14 after the end of the treatment
  Percentage of antibiotics prescribed, Choice of antibiotic class, whether 'delayed' or immediate, duration, posology

CONTACTS AND LOCATIONS:
Overall Officials: Véronique ORCEL, Dr, Principal Investigator — Département Universitaire d'Enseignement et de Recherche de Médecine Générale de Créteil
Locations (1):
- Cabinet de groupe, Saint-Maur-des-Fossés, Saint Maur, France

REFERENCES:
- [Background] Caron F, Galperine T, Flateau C, Azria R, Bonacorsi S, Bruyere F, Cariou G, Clouqueur E, Cohen R, Doco-Lecompte T, Elefant E, Faure K, Gauzit R, Gavazzi G, Lemaitre L, Raymond J, Senneville E, Sotto A, Subtil D, Trivalle C, Merens A, Etienne M. Practice guidelines for the management of adult community-acquired urinary tract infections. Med Mal Infect. 2018 Aug;48(5):327-358. doi: 10.1016/j.medmal.2018.03.005. Epub 2018 May 16. No abstract available. PMID 29759852
- [Background] Grigoryan L, Trautner BW, Gupta K. Diagnosis and management of urinary tract infections in the outpatient setting: a review. JAMA. 2014 Oct 22-29;312(16):1677-84. doi: 10.1001/jama.2014.12842. PMID 25335150
- [Background] Soudais B, Lacroix-Hugues V, Meunier F, Gillibert A, Darmon D, Schuers M. Diagnosis and management of male urinary tract infections: a need for new guidelines. Study from a French general practice electronic database. Fam Pract. 2021 Jul 28;38(4):432-440. doi: 10.1093/fampra/cmaa136. PMID 33340317
- [Background] Kinouani S, de Lary de Latour H, Joseph JP, Letrilliart L. Diagnostic strategies for urinary tract infections in French general practice. Med Mal Infect. 2017 Oct;47(6):401-408. doi: 10.1016/j.medmal.2017.05.003. Epub 2017 Jun 9. PMID 28606664
- [Background] Vincent YM, Frachon A, Buffeteau C, Conort G. Construction of a patient decision aid for the treatment of uncomplicated urinary tract infection in primary care. BMC Fam Pract. 2021 Jan 26;22(1):26. doi: 10.1186/s12875-021-01374-3. PMID 33499824
- [Background] Piraux A, Faure S, Naber KG, Alidjanov JF, Ramond-Roquin A. Changes in the management of urinary tract infections in women: impact of the new recommendations on antibiotic prescribing behavior in France, between 2014 and 2019. BMC Health Serv Res. 2021 Jun 28;21(1):612. doi: 10.1186/s12913-021-06653-4. PMID 34182991
- [Background] Lugtenberg M, Burgers JS, Zegers-van Schaick JM, Westert GP. Guidelines on uncomplicated urinary tract infections are difficult to follow: perceived barriers and suggested interventions. BMC Fam Pract. 2010 Jun 28;11:51. doi: 10.1186/1471-2296-11-51. PMID 20584276